CLINICAL TRIAL: NCT04853082
Title: Clinical Trial of Limonene on Regulating Metabolism-related Fatty Liver Disease (MAFLD) and Analysis of TCM Constitution
Brief Title: Limonene on Regulating Metabolism-related Fatty Liver Disease (MAFLD) and Analysis of TCM Constitution
Acronym: DL-MAFLD-TCM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hongsheng Tan (Other)
Collaborators: Shanghai Shen Kang Hospital Development Center (Other); Longhua Hospital (Other); Hongqiao International Institute of Medicine, Shanghai Tongren Hospital and Faculty of Public Health, Shanghai Jiao Tong University School of Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Hongsheng Tan, Associate Professor, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DL-MAFLD-TCM; SHDC2020CR4095 (Other Grant/Funding Number: Clinical Research Plan of SHDC)
Record Dates: First submitted 2021-04-05; First posted 2021-04-21 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Fatty Liver
Keywords: Metabolic associated fatty liver disease (MAFLD); Limonene; Efficacy; Safety
MeSH Terms: conditions — Fatty Liver | interventions — Limonene

STUDY DESIGN:
Intervention Model Description: Exploratory Clinical Trial；Randomized Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limonene capsules(marketed product in China) (Active Comparator): Limonene capsules(marketed product in China) donate by pharmaceutical company
  Interventions: Drug: Limonene capsule
- Limonene capsules(Placebo) (Placebo Comparator): Same smell, color and shape as limonene capsules(marketed product in China), without limonene in capsules
  Interventions: Drug: Limonene capsules(Placebo)

INTERVENTIONS:
Drug: Limonene capsule — All the recruiters will be given treatment under the guidance of basic diet. Basic dietary guidelines include high-quality protein and fresh green leafy vegetables. It need to controlled sugar, various sweets and high-calorie foods, frying and other foods with high oil content and foods with high cholesterol content. Limonene capsules group and placebo group were used for treatment. The random number is generated by the central randomization system. All the recruiters were divided into placebo control group and limonene capsule administration group. The numbers will be assigned according to random numbers. In this study, qualified subjects were randomly assigned to the treatment group and the placebo control group at a ratio of 1:1. The drug was administered for 12 weeks, 3 times a day, 5 capsules each time.
  Other Names: DAN LENING capsule
  Arms: Limonene capsules(marketed product in China)
Drug: Limonene capsules(Placebo) — Limonene capsules(Placebo)
  Arms: Limonene capsules(Placebo)

SUMMARY:
The prevention and treatment of metabolic-related fatty liver disease (MAFLD) involves many fields in preventive medicine and clinical medicine. So far, western medicine has not yet completed the elucidation of the mechanism of this type of disease, and there is a lack of effective therapeutic drugs.The purpose of this study was to evaluate the effectiveness and safety of limonene capsules (marketed product in China) in the treatment of metabolic-related fatty liver disease and related lipid-lowering mechanisms.

DETAILED DESCRIPTION:
In April 2020, in the famous journal "Journal of Hepatology" in the field of liver disease, an internationally renowned liver disease expert group jointly proposed to replace non-alcoholic fatty liver disease (NAFLD) with metabolic associated fatty liver disease (MAFLD) . The concept of non-alcoholic fatty liver disease (NAFLD) was first proposed by Ludwig in 1980. It specifically refers to the excessive deposition of liver fat without excessive drinking. It is a type of liver that is closely related to insulin resistance and genetic susceptibility. Non-alcoholic fatty liver disease (NAFLD) is China country's largest chronic liver disease and the primary cause of abnormal liver enzymes in health examinations. It can lead to liver disability and death. It is also closely related to a variety of metabolic diseases and the high incidence of colorectal tumors. Western medicine has not yet fully elucidated its mechanism, and no drugs have been officially approved for the clinical treatment of NAFLD.

The new MAFLD nomenclature highlights the central role of metabolic factors in causing liver fat deposition in this type of liver disease. Traditional Chinese medicine believes that the abnormal accumulation of fat in the liver of such fatty liver patients is a pathological product of the microscopic loss of water and valley essence. It belongs to phlegm stasis, which blocks the liver collaterals. It coincides with the core of the metabolic etiology of recent liver disease experts.

Limonene is widely found in the essential oils of traditional Chinese medicine tangerine peel, green peel and other plants. Its taste is sour, sweet and pungent.It is returned to the liver and gallbladder meridian. It has an aromatic odor effect.

A large number of animal and cell experiments in the early stage have shown that limonene can inhibit the differentiation of adipocytes (pre-adipocytes) and promote the apoptosis of mature adipocytes, which is related to the inhibition of fatty acid synthesis. Toxicity load experiments show that limonene has very low toxicity. The accumulation of lipids in the liver of mice has a regulatory effect with significantly reducing the content of liver cholesterol and triglycerides, and also has a certain effect on lipid metabolism disorders, hyperglycemia and other metabolic syndromes. It can alleviate the effects of high-fat diet and N- Efficacy of nitro-L-arginine methyl ester-induced resistance to non-alcoholic fatty liver in rats. The main indication of limonene capsules (marketed product in China) is liver and gallbladder diseases. Traditional Chinese medicine believes that liver and gallbladder are related to each other. This comprehensively shows that limonene capsules are promising to be developed as a pure Chinese medicine product for the safe and effective treatment of MAFLD.

However, there has been no clinical evaluation of the clinical efficacy of limonene in the treatment of metabolic-related fatty liver disease. As a typical aromatic Chinese medicine, the mechanism of limonene in the treatment of fatty liver urgently needs to be revealed by modern medicine and molecular biology techniques.

This study intends to use a randomized, double-blind, placebo-controlled method to evaluate the effect of limonene on improving the degree of fat infiltration in patients with metabolic-related fatty liver disease (MAFLD), and to evaluate its body mass index BMI, waist circumference, waist-to-hip ratio, subcutaneous fat thickness, fat percentage, changes in metabolic components, safety,etc. The study also intends to use metabonomics, genomics, and molecular biology techniques to study the clinical relationship between metabolites and physiological and pathological changes in patients with liver fat infiltration, and to detect changes in key proteins and lipid components after drug intervention, which is to reveal mechanism on treatment of metabolic-related fatty liver disease by limonene. It is aimed to study the difference in the efficacy of limonene for people with different constitutions of traditional Chinese medicine (TCM) combined with the analysis of the constitution of TCM, and to clarify the modern scientific attributes of TCM therapy. Finally the study will develop a safe and efficient drug treatment technology to control liver fat infiltration , and to promote the development of clinical disciplines in the treatment of metabolic-related fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis and imaging diagnosis of MAFLD and BMI index greater than or equal to 23kg/m2；
2. The age of the recruiter is between 18-65 years old;
3. Those who can cooperate with various treatments and data measurements according to the treatment cycle, and can persist in completing the test;
4. Those who accept and are willing to sign the informed consent.

Exclusion Criteria:

Potential recruiters who meet the inclusion criteria will be excluded if they meet any of the following:

1. Those who routinely take prescription drugs (except regular contraceptive drugs) or those who use auxiliary Chinese and Western drugs to treat non-alcoholic fatty liver;
2. Patients suffering from viral hepatitis, autoimmune hepatitis, hepatolenticular degeneration, hypothyroidism, infection, and biliary tract diseases that lead to abnormal liver function;
3. Patients who have taken the following drugs in the past 4 weeks: hypoglycemic drugs, lipid-lowering drugs (such as statins, fibrates, etc.) and drugs that may affect liver fat content (such as: silybin, ursodeoxycholic acid) , Bicyclic alcohol, phosphatidylcholine and vitamin E, glucocorticoid);
4. Patients with diabetes or those who have undergone bariatric surgery;
5. People who have gained or lost weight by 10 kg or more in the past two months;
6. People who are allergic to limonene capsules; or people who are allergic to citrus foods; people who especially like to eat a lot of citrus foods (daily dosage more than 100 grams);
7. Patients with severe cardiac insufficiency and malignant tumors;
8. Patients who have a history of mental illness and cannot cooperate with this project;
9. Pregnant and lactating women, or women or men who are willing to become pregnant or give birth during the study;
10. Participate in any other clinical trials;
11. Other situations where the researcher thinks it is inappropriate to participate in this research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Difference of controlled attenuation parameter (CAP) in liver fat | at baseline and twelve weeks after administration
  Changes in controlled attenuation parameter (CAP) in liver fat measured with transient elastography between the drug group and the placebo group.
Difference of rate of BMI index | at baseline, four, twelve weeks after administration
  The percent change of BMI index between the drug group and the placebo group.

SECONDARY OUTCOMES:
Difference of waist circumference | at baseline, four, twelve weeks after administration
  The percent change of waist circumference between the drug group and the placebo group.
Difference of aspartate transaminase (AST) index | at baseline, four, twelve weeks after administration
  The absolute values of changes in the levels of AST was compared between the two groups. Serum AST content of the patients were detected by an automatic biochemical analyzer before and after treatment.
Difference of glutamic transpeptidase (GGT) index | at baseline, four, twelve weeks after administration
  The absolute values of changes in the levels of GGT was compared between the two groups. Serum GGT content of the patients were detected by an automatic biochemical analyzer before and after treatment.
Difference of alanine transaminase (ALT) index | at baseline, four, twelve weeks after administration
  The absolute values of changes in the levels of ALT was compared between the two groups. Serum ALT content of the patients were detected by an automatic biochemical analyzer before and after treatment.
Difference of total cholesterol (TC) index | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of TC was compared between the two groups before and after treatment. Serum TC content of the patients were detected by an automatic biochemical analyzer before and after treatment.
Difference of glycerin trilaurate (TG) index | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of TG was compared between the two groups before and after treatment. Serum TG content of the patients were detected by an automatic biochemical analyzer before and after treatment.
Difference of low-density lipoprotein cholesterol (LDL-C) index | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of LDLC was compared between the two groups before and after treatment. Serum LDL-C content of the patients were detected by an automatic biochemical analyzer before and after treatment.
Difference of high-density liptein cholesterol（HDL-C）index | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of HDL-C was compared between the two groups before and after treatment. Serum HDL-C content of the patients were detected by an automatic biochemical analyzer before and after treatment.
Difference of apolipoprotein E (ApoE) index | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of ApoE was compared between the two groups before and after treatment. Serum ApoE content of the patients were detected by an automatic biochemical analyzer before and after treatment.
Difference of insulin index | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of insulin was compared between the two groups before and after treatment.
Difference of glycated hemoglobin（GHb）index | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of GHb was compared between the two groups before and after treatment.
Difference of blood sugar index | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of blood sugar was compared between the two groups before and after treatment.
Difference of the Short Form 36 physical component summary (SF-36 PCS) score | at baseline, two，four，six，eight，ten weeks, twelve and sixteen weeks after administration
  Using the Telephone Interview for the SF-36 PCS score (range, 0 [worst] to 100 [best]).
Difference of the Chronic Liver Disease Questionnaire (CLDQ) | at baseline, two，four，six，eight，ten weeks, twelve and sixteen weeks after administration
  Using the Telephone Interview for the CLDQ score (range, 0 [worst] to 100 [best]).
Difference of the Traditional Chinese of Medicine ( TCM ) Physique Questionnaire | at baseline, two，four，six，eight，ten weeks, twelve and sixteen weeks after administration
  Using the Telephone Interview for the TCM Physique Questionnaire score (range, 0 [worst] to 100 [best]).

OTHER OUTCOMES:
Difference of CRP related to the mechanism of action | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of CRP were compared between the two groups before and after treatment.
Difference of IL6 related to the mechanism of action | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of IL6 were compared between the two groups before and after treatment.
Difference of TNF-a related to the mechanism of action | at baseline, twelve weeks after administration
  The absolute values of changes in the levels of TNF-a were compared between the two groups before and after treatment.
Difference of lipidomics metabolites of blood | at baseline, twelve weeks after administration
  The metabolomics and genomics detection methods of ultra-high performance liquid chromatography combined with quadrupole time-of-flight mass spectrometry (UPLC-QTOF-MS) were used to test the serum lipid compounds of all samples. Collect 5 mL of fasting venous blood from the subjects in the morning. Obtain serum samples after centrifugation. And then perform lipidomics test.
Adverse Events | sixteen weeks
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Qian, Doctor, Principal Investigator — Shanghai Shen Kang Hospital Development Center;Hongqiao International Institute of Medicine, Shanghai Tongren Hospital and Faculty of Public Health, Shanghai Jiao Tong University School of Medicine; Xiaoyun Chen, Doctor, Principal Investigator — Longhua Hospital; Hongsheng Tan, Doctor, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Longhua Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Eslam M, Newsome PN, Sarin SK, Anstee QM, Targher G, Romero-Gomez M, Zelber-Sagi S, Wai-Sun Wong V, Dufour JF, Schattenberg JM, Kawaguchi T, Arrese M, Valenti L, Shiha G, Tiribelli C, Yki-Jarvinen H, Fan JG, Gronbaek H, Yilmaz Y, Cortez-Pinto H, Oliveira CP, Bedossa P, Adams LA, Zheng MH, Fouad Y, Chan WK, Mendez-Sanchez N, Ahn SH, Castera L, Bugianesi E, Ratziu V, George J. A new definition for metabolic dysfunction-associated fatty liver disease: An international expert consensus statement. J Hepatol. 2020 Jul;73(1):202-209. doi: 10.1016/j.jhep.2020.03.039. Epub 2020 Apr 8. PMID 32278004